CLINICAL TRIAL: NCT00621673
Title: Assessment of the Risk of Inhibitor Formation in Subjects With Severe Hemophilia A When Switched From a Replacement Therapy With a rFVIII Produced by a Chinese Hamster Ovary (CHO) Cell Line to a rFVIII Produced by a Baby Hamster Kidney (BHK) Cell Line (Kogenate® FS).
Brief Title: Assessment of the Risk of Inhibitor Formation in Previously Treated Patients With Severe Hemophilia A
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 12112
Record Dates: First submitted 2008-02-12; First posted 2008-02-22 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Hemophilia A
Keywords: Hemophilia A,; Inhibitor formation,; rFVIII
MeSH Terms: conditions — Hemophilia A | interventions — F8 protein, human; BAY 14-2222

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Drug: Kogenate (BAY 14-2222)

INTERVENTIONS:
Drug: Kogenate (BAY 14-2222) — Antihemophilic factor (recombinant) 20-40 IU/ kg based on body weight of rFVIII, IV, 3 times a week

SUMMARY:
Most transient inhibitor formation, if any, will develop within the first 4 weeks. The study is to further monitor whether participants with severe Hemophilia A will develop inhibitors or antibodies at the later stage when switched from their current recombinant therapy produced from Chinese Hamster Ovary (CHO) cell line to Kogenate-FS raised in a Baby Hamster Kidney cell line.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with severe hemophilia A (< 2% FVIII:C)
* Subjects with no history of FVIII inhibitor antibody formation
* Subjects with no measurable inhibitor activity
* Subjects with at least 200 EDs with FVIII concentrate in total, including 20 EDs in the previous 6 months
* Subjects whose current treatment with any CHO rFVIII product
* Subjects with no elective surgery and/or continuous infusion FVIII administration is foreseen during the study
* Subjects with normal prothrombin time (PT), partial thromboplastin time (PTT) compatible with FVIII deficiency

Exclusion Criteria:

* Subjects with any other bleeding disease beside hemophilia A (i,e., von Willebrand's disease)
* Subjects who have known intolerance or allergic reactions to constituents of rFVIII-FS or known hypersensitivity to mouse or hamster proteins
* Any individual with a past history of severe reaction(s) to FVIII concentrates
* Subjects on treatment with immunomodulatory agents within the last 3 months prior to study entry
* Subjects who were receiving or had received other experimental drugs within 3 months prior to study entry
* Subjects who require any medication for FVIII infusions

Ages: 12 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2006-05; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
To evaluate whether a switch of replacement therapy from an rFVIII produced in a CHO cell line to an rFVIII produced in a BHK cell line is associated with a risk of inhibitor formation. | 6 months

SECONDARY OUTCOMES:
To quantify the risk of inhibitor formation, to assess the efficacy of the rFVIII-FS while on regular replacement therapy and to assess the quality-of-life (QoL) before and after the study. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (2):
- United States (2):
  - Detroit, Michigan
  - Las Vegas, Nevada